CLINICAL TRIAL: NCT03553472
Title: Identify Young Immunosuppressed and Non-immunosuppressed Inflammatory Bowel Disease Patients at Risk for HZ
Brief Title: Identifying Young Inflammatory Bowel Disease Patients at Risk for Herpes Zoster
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0512
Record Dates: First submitted 2018-01-22; First posted 2018-06-12 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Herpes Zoster; Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Herpes Zoster; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — ELISPOT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Non-immunosuppressed IBD patients: 24 IBD patients on mesalamine therapy or no IBD therapy
- Thiopurine group: 12 IBD patients on azathioprine at least 2.0mg/kg or 6MP 1.0mg/kg
- Anti-TNF therapy: 12 IBD patients on maintenance therapy infliximab (at least 8 every 8 weeks), golilumab (at least monthly), adalilumab (at least every 2 weeks), or certolizumab (at least monthly)
- Combination therapy: 12 IBD patients on anti-TNF therapy as described in group along with either 15mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg
- Healthy Control: The control group with consist of 12 individuals who meet the following inclusion and exclusion criteria.
  Individuals will be obtained from patients without an IBD diagnosis, chronic liver disease, celiac disease or other chronic health condition coming to Digestive Health Center for endoscopic procedures or clinic visits.
- Vedolizumab therarpy: 12 IBD patients on vedolizumab maintenance therapy every 4-8 weeks
- Prednisone and Anti-TNF therapy: 12 IBD patients on Anti-TNF maintenance therapy as combination or mono therapy along with at least 10mg of prednisone

SUMMARY:
Inflammatory bowel disease (IBD) patients under the age of 50 can have a greater risk than the general population above age 50. IBD patient are commonly treated with immunosuppression that increases the risk for Herpes Zoster. A new HZ vaccine is available that could decrease the risk of HZ in IBD patients.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a group of chronic inflammatory disorders of the gastrointestinal tract. A recent national survey from the CDC estimates that the prevalence of IBD in the United States (US) is nearly 3.1 million cases. IBD is often associated with debilitating symptoms, hospitalizations, decreased quality of life, frequent procedures and/or surgery. Treatment options include immunosuppressive therapies, such as corticosteroids, immunomodulators (thiopurines and methotrexate) and anti-tumor necrosis factor alpha (TNF) agents. Although they are effective in achieving clinical remission and decrease the risk of complications, they also increase the risk for serious infections, including herpes zoster (HZ).

The primary goal is to study those patients with IBD who are thought to be at the highest risk for HZ reactivation by evaluating cell mediated immunity (CMI) to VZV.

ELIGIBILITY:
Inclusion Criteria:

A history of chronic (greater than 3 month) ulcerative colitis or Crohn's disease diagnosed and documented by the standard clinical, radiographic, endoscopic and histopathologic criteria.

3.12 Ages 40-55 3.13 There will four groups divided by medication group. All patients will be on stable doses of medication for at least 3 months divided in the following groups: A) Group A (24 patients): mesalamine therapy or no IBD therapy B) Group B (12 patients): Thiopurine group: On azathiopurine at least 2.0mg/kg or 6MP 1.0mg/kg C) Group C (12 patients): Anti-TNF therapy group: On maintenance therapy infliximab (at least 8 every 8 weeks), golilumab (at least monthly), adalilumab (at least every 2 weeks), or certolizumab (at least monthly) D) Group D (12 patients): Combination therapy: On anti-TNF therapy as described in group along with either 15mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg 3.14 Previous history of varicella infection verified by positive VZV IgG test. 3.15 The patient must understand and voluntarily sign the informed consent document.

3.16 All participants must have received a tetanus, diphtheria, pertussis (Tdap) or tetanus, diphtheria (Td) within the previous 10 years the Wisconsin Immunization Registry (WIR), will be accessed via the EMR, so confirming immunization will not be a limitation) because tetanus CMI will be used as an experimental control.

Exclusion Criteria:

3.21 Current use of systemic steroids 3.22 Other autoimmune condition (e.g Rheumatoid arthritis, autoimmune hepatitis) 3.23 Receipt of HZ vaccine (As above, via WIR) 3.24 History of cytopenia in the last 12 months (WBC < 3.0 or anemia Hgb <10). (All patients on immunosuppressants routinely obtain blood work every 3-6 months, so this will be available at study entry) 3.25 History of previous herpes zoster infection.

Ages: 35 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: IBD patients with confirmed IBD
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Immune response by T cell, cell mediated immunity, to varicella zoster virus in patients with inflammatory bowel disease. | Day 1
  ELISPOT is an enzyme-linked assay for detecting and enumerating cytokine-producing lymphocytes. ELISPOT can detect cytokine-producing cells in as few as 1 in 300,000 cells. ELISPOT is the standard for measuring varicella cell mediated immunity.

SECONDARY OUTCOMES:
Immune response by T cells ,cell Mediated Immunity, to varicella zoster virus in Immunosuppressed patients with IBD compared to those non-Immunosuppressed | Day 1
  ELISPOT is an enzyme-linked assay for detecting and enumerating cytokine-producing lymphocytes. ELISPOT can detect cytokine-producing cells in as few as 1 in 300,000 cells. ELISPOT is the standard for measuring varicella cell mediated immunity.
Immune response by T cell, cell mediated immunity, to varicella zoster virus in Immunosuppressed IBD patients compared to other immunosuppressed IBD patients | Day 1
  ELISPOT is an enzyme-linked assay for detecting and enumerating cytokine-producing lymphocytes. ELISPOT can detect cytokine-producing cells in as few as 1 in 300,000 cells. ELISPOT is the standard for measuring varicella .

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Caldera, DO, Principal Investigator — University of Wisconsin School of Medicine
Locations (1):
- University of Wisconsin Digestive Health Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided